CLINICAL TRIAL: NCT03182517
Title: Correlation of Parathyroid Hyperplasia by Ultrasound With Clinical and Laboratory Findings in Patients With Chronic Kidney Disease.
Brief Title: Parathyroid Hyperplasia in Patients With Chronic Kidney Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: PTH
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic kidney diseases: patients with chronic renal failure on dialysis since 3-5 years

SUMMARY:
Secondary hyperparathyroidism is an important complication in patient with chronic kidney disease . It is associated with bone complication and an increase in cardiovascular mortality The parathyroid hormone rises in these patients as consequence of low concentration of vitamin D3 ,reduction in quantities of serum calcium, phosphorus retention and reduction of vitamin D receptors sensitive to calcium.

ELIGIBILITY:
Inclusion Criteria:

* stage 5 chronic renal failure
* dialysis (peritoneal ,or hemodialysis) since 3---5 years

Exclusion Criteria:

* previous of neck surgery.
* Patients refusal to participate in the study or voluntary withdrawal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic renal diseases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with high parathyroid hormone level | 1 day
  laboratory measurement of parathyroid hormone

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No